CLINICAL TRIAL: NCT00777933
Title: Randomized Trial of Cyclosporine and Tacrolimus Therapy With Steroid Withdrawal in Living-Donor Renal Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Jae-Won Joh, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000-07-02
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Kidney Transplantation; Living Donors
MeSH Terms: interventions — Tacrolimus; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cyclosporine (Active Comparator)
  Interventions: Drug: cyclosporine
- Tacrolimus (Experimental)
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: tacrolimus
  Arms: Tacrolimus
Drug: cyclosporine
  Arms: cyclosporine

SUMMARY:
The use of steroids after kidney transplantation has been challenged because of variable adverse effects which may increase the patient morbidity and mortality. The aim of this study was to compare the safety and efficacy of immunosuppressive regimens consisting of cyclosporine (CsA) and mycophenolate mofetil (MMF) or tacrolimus (TAC) and MMF after steroid withdrawal 6 months after kidney transplantation in low-risk patients.

DETAILED DESCRIPTION:
131 patients were randomized to CsA (n = 63) or TAC (n = 68). Of 118 patients who did not have a biopsy-proven rejection episode and who had a serum creatinine level < 2.0 mg/dL 6 months after transplantation, 55 were of the CsA group and 63 were of the TAC group. We assessed patient and graft survival, acute rejection episodes, and adverse events 5 years after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* older than 15 years
* first living donor kidney transplantation

Exclusion Criteria:

* congestive heart failure (ejection fraction < 35%)
* chronic liver disease
* underlying diabetes mellitus
* evidence of systemic infection at screening time
* history of malignant disease
* multiple organ transplantation
* positive serologic evidence of human immunodeficiency virus

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2000-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Graft survival | 5 years
Patient survival | 5 years

SECONDARY OUTCOMES:
cumulative incidence of acute rejection | 5 years
estimated glomerular filtration rate | 5 year
new-onset diabetes mellitus | 5 year
Hypertension | 5 year
hyperlipidemia | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Won Joh, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Transplantation Center, Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee YJ, Kim B, Lee JE, Kim YG, Kim DJ, Kim SJ, Joh JW, Oh HY, Huh W. Randomized trial of cyclosporine and tacrolimus therapy with steroid withdrawal in living-donor renal transplantation: 5-year follow-up. Transpl Int. 2010 Feb;23(2):147-54. doi: 10.1111/j.1432-2277.2009.00955.x. Epub 2009 Sep 9. PMID 19744223